CLINICAL TRIAL: NCT02044133
Title: Monocentric Randomized Study, Assessing the Interests of the Determination of Vitamin D in Prison Population. (Vitamine D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHD026-12
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Male Prisoner

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dosage of vitamine D : inclusion and 6 month (Other): Participant will have one dosage of vitamine D to entrance of prison and one dosage of vitamine D 6 month after entry
  Interventions: Other: Dosage Vitamine D
- Dosage of Vitamine D 6 month (Other): Participant will have one dosage of vitamine D 6 month after entry to prison
  Interventions: Other: Dosage Vitamine D

INTERVENTIONS:
Other: Dosage Vitamine D

SUMMARY:
The study will be proposed to man entering the prison of La Roche sur Yon. Participants will be randomized into two arms: one arm realize a dosage of vitamin D at the entrance and 6 months after the entry and the second arm will carry only a dosage six months after entry.

the purpose of the study is to determine the interest of dosage of vitamin D in biological assessment of entry into prison house.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated person
* Imprisoned in La Roche sur Yon
* Male
* Age > 18 year old
* Not opposed to participation in the study

Exclusion Criteria:

* Intellectual deficit not to understand the study
* Taking osteoporosis treatment or any other affecting the metabolism of vitamin D
* Renal failure, liver failure
* Hypercalcemia
* Thyroid dysfunction, parathyroid diseases
* Duration of imprisonment less than the expected duration of the study.
* Incarcerated person who had received supplementation of vitamin D in the 6 months prior

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves BLEHER, PH, Principal Investigator — CHD Vendée La Roche sur Yon
Locations (1):
- Centre hospitalier départemental Vendée, La Roche-sur-Yon, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruted based on physicien referral between september 2013 and january 2016. The first participant was enrolled on january 29, 2014 and the last participant was enrolled in july 15, 2015. 54 patients met inclusion criteria and were randomized.
Groups:
- Dosage of Vitamine D : Inclusion and 6 Month: Participant will have one dosage of vitamine D to entrance of prison and one dosage of vitamine D 6 month after entry
  Dosage Vitamine D
- Dosage of Vitamine D 6 Month: Participant will have one dosage of vitamine D 6 month after entry to prison
  Dosage Vitamine D
Period: Overall Study
Arm/Group | Dosage of Vitamine D : Inclusion and 6 Month | Dosage of Vitamine D 6 Month
Started | 26 | 28
Completed | 20 | 22
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 1 | 0
Not completed — Release | 3 | 4
Not completed — Transfer | 1 | 0
Not completed — refusal of blood sampling | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dosage of Vitamine D : Inclusion and 6 Month | Dosage of Vitamine D 6 Month | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (8.5) | 35.3 (11.9) | 32.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 28 | 54
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Dosage of Vitamin D
Description: Vitamin D level in ng/mL
Time Frame: 6 month
Population: ITT analyse
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dosage of Vitamine D : Inclusion and 6 Month | Dosage of Vitamine D 6 Month
Number analyzed (Participants) | 26 | 28
ng/mL | 28.2 (8.6) | 14.6 (9.8)
Statistical Analysis 1: Comparison: Dosage of Vitamine D : Inclusion and 6 Month vs Dosage of Vitamine D 6 Month; Test type: Superiority; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: The planned follow-up period for patients is six months until the M6 visit.
Arm/Group | Dosage of Vitamine D : Inclusion and 6 Month | Dosage of Vitamine D 6 Month
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 0/26 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes